CLINICAL TRIAL: NCT01853423
Title: Tuberous Sclerosis Complex: Facial Angiofibroma Skin Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Le Bonheur Children's Hospital (Other)
Collaborators: Pfizer (Industry); University of Tennessee (Other)
Responsible Party: Principal Investigator, James W. Wheless, Medical Doctor, Le Bonheur Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTHSC TSC01; 12-2008 (Other: Instututional Review Board)
Record Dates: First submitted 2013-04-12; First posted 2013-05-15 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Facial Angiofibroma
Keywords: Rapamune; Topical; Pediatric; Safety; Efficiency; Angiofibroma; Skin Cream
MeSH Terms: conditions — Tuberous Sclerosis; Angiofibroma | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rapamune (Experimental): Small amount of 0.1% rapamune ointment applied topically to affected facial areas twice daily for the first two weeks, then once daily.
  Interventions: Drug: Rapamune

INTERVENTIONS:
Drug: Rapamune — Small amount of 0.1% rapamune ointment applied topically to affected facial areas twice daily for the first two weeks, then once daily.
  Other Names: Sirolimus

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of a 0.1% formulation of rapamune cream in children with Tuberous Sclerosis Complex (TSC), ages 3 years and older, who have facial angiofibromas that would benefit from treatment.

DETAILED DESCRIPTION:
This is an open label, prospective single center study. Patients that are seen in our regional Tuberous Sclerosis Complex Clinic and have facial angiofibromas that would benefit from this cream and who wish to be involved in this study would be enrolled. We anticipate enrolling 12-15 patients the first year. Patients will have pictures of their facial angiofibromas taken immediately prior to entry into the study. They will then be prescribed 0.1% rapamune topical formulation to apply twice daily to their skin for the first two weeks and then once daily. If level is above 0, will re-check serum lipids, cbc, and repeat levels every three-four months and monitor the patient for symptoms. Patients will return at one month and three months to obtain serum rapamune levels along with pictures, then they will be seen intermittently throughout the first year with photographs of their face taken at the one month visit, 3 month visit, six month visit and twelve month visit. We will ask the parents about any side effects from the medication during the entire time patients are using the topical rapamune. We will monitor the facial lesions as well. We will assess for skin sensitivity, pain, erythema, or pruritus. If skin irritation results from the drug, then we will stop use of the drug. Parents will sign an informed consent allowing their child's picture to be taken and allowing us to summarize the data for publication at the end of this study.

This study will be the first study using a consistent formulation to make a 0.1% rapamune cream, and this will be performed under the direction of myself and Dr. Almoazen in the University of Tennessee Health Science Center(UTHSC) College of Pharmacy compounding laboratory. Only patients who are thought to be reliable for the follow up visits and to use the cream appropriately will be enrolled in the study. This study meets the FDA criteria for an Investigational New Drug(IND) exemption.

The adverse events noted in the package insert for rapamune cream are all based on systemic administration of the medication, primarily to adults with other diseases. In our clinical experience, with topical use there is no absorption and we have not noted any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient or his / her legally authorize representative (LAR) must sign and date the approved informed consent prior to study participation or initiation of study procedures. If appropriate, the patient will give written or verbal consent. Surrogate consent will be obtained utilizing the "legally authorized representative (LAR)". The LAR must be an adult who has exhibited special care and concern for the subject, who is familiar with the subject's personal values, who is reasonably available, and who is willing to serve. No person who is identified as a protective order or other court order that directs that person to avoid contact with the subject shall be eligible to serve as the subject's LAR. Identification of LAR should normally be made using the following order of descending preference: Conservator, guardian, attorney in fact, subject's spouse (unless legally separated), the subject's adult child, the subject's parent, the subject's adult sibling, any other adult relative of the subject, or other adult who is familiar with the patient's personal values, who is reasonably available, and who is willing to serve.

  1. Patient must have a diagnosis of Tuberous Sclerosis Complex.
  2. Female or male patients over the age of 3 years.
  3. Female subjects of child bearing potential must not be pregnant and must undergo a pregnancy test, and must agree to use appropriate contraceptive methods

     Exclusion Criteria:
* Patients will be excluded from entry into the study if any of the following are true:

  1. Patient has a history of drug allergy to rapamune.
  2. Patient is pregnant or lactating.
  3. Subject is receiving therapy with Rapamycin.
  4. Subject is receiving any form of immunosuppression or has previously experienced immune dysfunction.
  5. Subject is currently participating in or has participated within the Last 30 days in a clinical trial involving an investigative drug.
  6. Subject has other dermatologic conditions that would preclude or prevent adequate assessment of changes to their facial angiofibromas.
  7. Subject has had laser surgery, cryotherapy, or other dermatologic treatment to their facial angiofibromas within the previous 6 months.

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2013-10; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Reduction of facial angiofibroma with use of rapamune facial skin cream | 1 year
  1. Tolerability: Number of participants with adverse events
  2. Efficacy: Skin assessment to measure improvement of facial angiofibromas
  3. Safety: Rapamune levels (serum)

CONTACTS AND LOCATIONS:
Overall Officials: James W Wheless, MD, Principal Investigator — LeBonheur Children's Hospital- Neuroscience Institute
Locations (1):
- LeBonheur Children's Hospital, Memphis, Tennessee, United States